CLINICAL TRIAL: NCT02324712
Title: Cytokine and Growth Factor Changes and Correlation With Clinical Outcomes Following Acupuncture for TMD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI relocated to another institution; study may be resubmitted at a later date.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-0919
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Active Comparator): Acupuncture treatment for TMD
  Interventions: Device: Acupuncture
- Sham Acupuncture (Sham Comparator): Acupuncture treatment for TMD using the non-penetrating Park Sham Acupuncture Device
  Interventions: Device: Sham Acupuncture

INTERVENTIONS:
Device: Acupuncture — Acupuncture using standard stainless steel acupuncture needles inserted into intramuscular tissue for 20 minutes
  Arms: Acupuncture
Device: Sham Acupuncture — Acupuncture using non-penetrating Park Sham Needles for 20 minutes
  Arms: Sham Acupuncture

SUMMARY:
Purpose: 1) To investigate differences in pro-inflammatory and anti-inflammatory cytokines and growth factors in the circulating blood (and cytokine levels only in saliva) of patients with chronic temporomandibular disorder (TMD) before and after acupuncture; 2) To determine differences in cytokine profiles between real and sham acupuncture in circulating blood of patients with chronic TMD; and 3) To explore correlations between these changes and clinical outcomes.

Participants: Patients with chronic TMD pain recruited through the University of North Carolina-Chapel Hill (UNC-CH) Orofacial Pain Clinic.

Procedures (methods): Participants will complete a self-administered questionnaire assessing TMD-related comorbidity. During the initial visit, study examiners will record clinical characteristics of muscles and joints of the head, neck and body according to newly recommended diagnostic criteria (DC) for TMD. Clinical outcomes include a pain index (computed from numeric rating scales) of masseter, temporalis and the supplemental painful muscles, and patient-reported symptoms (using the Measure Yourself Medical Outcome Profile; MYMOP) and pain intensity (using the Pain Scale). Blood (5 cc) will be taken before and after acupuncture treatments. Participants will self-collect pre-treatment and post-treatment saliva samples. Patients will receive 4 acupuncture treatments, once per week for 4 weeks. The primary outcome measure is change in IL-8 levels in circulating blood and saliva after 4 weeks of real acupuncture compared with sham acupuncture. Secondary outcome measures include comparing changes in levels of nerve growth factor (NGF), tumor necrosis factor-alpha (TNFα),vascular endothelial growth factor (VEGF), platelet-derived growth factor (PDGF), basic fibroblast growth factor (bFGF), and IL-1α, IL-2, IL-4, IL-6 and IL-10, before and after real acupuncture at Week 1 compared with sham acupuncture and before and after real acupuncture at Week 4 compared with sham acupuncture. The exploratory outcome measure is correlation between changes in cytokine levels and clinical variables after 4 weeks of real acupuncture compared with 4 weeks of sham acupuncture.

DETAILED DESCRIPTION:
Temporomandibular disorder (TMD) is known to be the second most frequent musculoskeletal pain condition following low back pain. According to the NIDCR, TMD affects 5%-12% of the population at an annual cost estimated at 4 billion dollars in the US. Recent studies that have investigated acupuncture as a treatment for musculoskeletal pain have reported various results. Several meta-analyses and systematic reviews of randomized controlled trials suggest that acupuncture treatment improves TMD-related pain. Its mechanism of action in improving TMD pain, however, is largely unclear.

Elevated levels of pro-inflammatory cytokines, e.g., MCP-1 and IL-8 have been found in circulating blood of patients with TMD. Upregulated pro-inflammatory cytokine levels have been correlated with greater sensitivity to pain evoking stimuli. Abnormalities in levels of pro-inflammatory cytokines are often accompanied by alterations in levels of anti-inflammatory cytokines, e.g., IL-1ra, which are associated with reductions in pain and inflammation. The effects of acupuncture on pro- and anti-inflammatory cytokines, growth factors, and clinical pain and function have not been reported in a prospective cohort of TMD patients at multiple time points in the clinical setting. The proposed mechanistic study seeks to ascertain if acupuncture compared to sham acupuncture produces measurable changes in circulating pro- and anti-inflammatory cytokines and growth factors in a manner that is associated with patient self-reports of pain and function over a 4-week treatment period. Cytokine and growth factor levels will be measured in blood and saliva; saliva will be used to measure cytokine levels only.

ELIGIBILITY:
Inclusion Criteria:

Signed, informed consent; females and males aged 18-64; planning on living in the area for the next 2 months; fluent in written and spoken English;

Myofascial pain with referral diagnosed according to TMD diagnostic criteria (Schiffman et al. 2014):

pain in the temporalis and masseter muscles report of familiar pain with palpation of the two muscles report of pain at a site beyond the boundary of the muscle being palpated.

Exclusion Criteria:

Traumatic facial injury or surgery on the face or jaw; currently receiving orthodontic treatment;

Systemic inflammatory disorders such as lupus, kidney failure or renal dialysis, heart disease or heart failure, chronic respiratory disease, hypertension, un- controlled diabetes, epilepsy or seizures

Hyperthyroidism; chemotherapy or radiation therapy; trigeminal neuralgia; cluster headache;

Drug or alcohol abuse; active or uncontrolled psychiatric disorders or recent (within 6 months) psychiatric hospitalization; pending pension or worker's claim/litigation; previous experience with acupuncture for TMD

Current use of NSAIDS and/or steroidal medications.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in cytokine IL-8 levels in circulating blood and saliva after 4 weeks of real acupuncture compared with 4 weeks of sham acupuncture. | Baseline, 4 weeks

SECONDARY OUTCOMES:
Change in patient-reported symptoms on the Measure Yourself Medical Outcome Profile (MYMOP; a 1-page paper questionnaire) after 4 weeks of real acupuncture compared with 4 weeks of sham acupuncture. | Baseline, 4 weeks
Change in patient-reported pain intensity on the Pain Scale (a 1-page paper questionnaire) after 4 weeks of real acupuncture compared with 4 weeks of sham acupuncture. | Baseline, 4 weeks
Change in cytokine MCP-1 levels in circulating blood and saliva after 4 weeks of real acupuncture compared with 4 weeks of sham acupuncture. | Baseline, 4 weeks
Change in cytokine IL-1ra levels in circulating blood and saliva after 4 weeks of real acupuncture compared with 4 weeks of sham acupuncture. | Baseline, 4 weeks
Change in cytokine IL-2 levels in circulating blood and saliva prior to and after real acupuncture compared with sham acupuncture at study Week 1. | Week 1
Change in cytokine IL-4 levels in circulating blood and saliva prior to and after real acupuncture compared with sham acupuncture at study Week 1. | Week 1
Change in cytokine IL-6 levels in circulating blood and saliva prior to and after real acupuncture compared with sham acupuncture at study Week 1. | Week 1
Change in cytokine IL-10 levels in circulating blood and saliva prior to and after real acupuncture compared with sham acupuncture at study Week 1. | Week 1
Change in cytokine IL-2 levels in circulating blood and saliva prior to and after real acupuncture compared with sham acupuncture at study Week 4. | Week 4
Change in cytokine IL-4 levels in circulating blood and saliva prior to and after real acupuncture compared with sham acupuncture at study Week 4. | Week 4
Change in cytokine IL-6 levels in circulating blood and saliva prior to and after real acupuncture compared with sham acupuncture at study Week 4. | Week 4
Change in cytokine IL-10 levels in circulating blood and saliva prior to and after real acupuncture compared with sham acupuncture at study Week 4. | Week 4
Change in nerve growth factor (NGF) levels in circulating blood prior to and after real acupuncture compared with sham acupuncture at study Week 1. | Week 1
Change in vascular endothelial growth factor (VEGF) levels in circulating blood prior to and after real acupuncture compared with sham acupuncture at study Week 1. | Week 1
Change in platelet-derived growth factor (PDGF) levels in circulating blood prior to and after real acupuncture compared with sham acupuncture at study Week 1. | Week 1
Change in basic fibroblast growth factor (bFGF) levels in circulating blood prior to and after real acupuncture compared with sham acupuncture at study Week 1. | Week 1
Change in tumor necrosis factor alpha (TNFa) levels in circulating blood prior to and after real acupuncture compared with sham acupuncture at study Week 1. | Week 1
Change in nerve growth factor (NGF) levels in circulating blood prior to and after real acupuncture compared with sham acupuncture at study Week 4. | Week 4
Change in vascular endothelial growth factor (VEGF) levels in circulating blood prior to and after real acupuncture compared with sham acupuncture at study Week 4. | Week 4
Change in platelet-derived growth factor (PDGF) levels in circulating blood prior to and after real acupuncture compared with sham acupuncture at study Week 4. | Week 4
Change in basic fibroblast growth factor (bFGF) levels in circulating blood prior to and after real acupuncture compared with sham acupuncture at study Week 4. | Week 4
Change in tumor necrosis factor alpha (TNFa) levels in circulating blood prior to and after real acupuncture compared with sham acupuncture at study Week 4. | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Jongbae (Jay) Park, KMD, PhD, Principal Investigator — University of North Carolina, Chapel Hill

REFERENCES:
- [Background] Cho SH, Whang WW. Acupuncture for temporomandibular disorders: a systematic review. J Orofac Pain. 2010 Spring;24(2):152-62. PMID 20401353
- [Background] La Touche R, Goddard G, De-la-Hoz JL, Wang K, Paris-Alemany A, Angulo-Diaz-Parreno S, Mesa J, Hernandez M. Acupuncture in the treatment of pain in temporomandibular disorders: a systematic review and meta-analysis of randomized controlled trials. Clin J Pain. 2010 Jul-Aug;26(6):541-50. doi: 10.1097/AJP.0b013e3181e2697e. PMID 20551730
- [Background] Slade GD, Conrad MS, Diatchenko L, Rashid NU, Zhong S, Smith S, Rhodes J, Medvedev A, Makarov S, Maixner W, Nackley AG. Cytokine biomarkers and chronic pain: association of genes, transcription, and circulating proteins with temporomandibular disorders and widespread palpation tenderness. Pain. 2011 Dec;152(12):2802-2812. doi: 10.1016/j.pain.2011.09.005. Epub 2011 Oct 14. PMID 22000099